CLINICAL TRIAL: NCT06579547
Title: Single-center Prospective Comparison of Diagnostic Performance of Deep-learning Agumented UTE/ZTE MRI Sequences and Standard-of-care Low Dose CT for Rheumatologic Patients With Musculoskeletal Disease
Brief Title: Evaluating Replacement of Standard-of-care Low Dose Computer Tomography (CT) Scans With Radiation-free Bone Imaging by Deep-learning Augmented Zero Echo Time (DL-ZTE) Magnetic Resonance Tomography (MRT)
Acronym: DLZTECT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Roman Guggenberger (Other)
Responsible Party: Sponsor-Investigator, Roman Guggenberger, Senior Physician (Leitender Arzt), University of Zurich
Organization: University of Zurich (Other)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: DLZTECT
Record Dates: First submitted 2024-08-23; First posted 2024-08-30 (Actual); Last update posted 2024-08-30 (Actual); Status verified 2024-08

CONDITIONS: Joint Diseases; Joint Inflammation
MeSH Terms: conditions — Joint Diseases; Arthritis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiologists who perform the readout will be blinded to the reference low dose CT scan to avoid being primed for certain bony anatomy and pathology by evaluating the low dose CT first. The reference low dose CT scan will be read in a separate session.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: Low Dose Computer Tomography — Participants will undergo MRI scans of their skeletal system, followed by the Intervention of a Low Dose CT scan of the same body region for comparison purposes.

SUMMARY:
The goal of this clinical trial is to determine how effectively bone structures of the human skeleton can be visualized using Deep Learning (DL) augmented Magnetic Resonance Imaging (MRI) in individuals with inflammatory and degenerative joint changes, compared to Computed Tomography (CT). MRI is a technique that operates without the use of X-rays. The main question it aims to answer is:

1. Can DL MRI accurately depict bone structures as well as CT?
2. Can DL MRI be used as an alternative to CT to avoid exposure to X-rays in the future?

Researchers will compare DL MRI scans to CT scans to see if DL MRI can effectively replace CT in visualizing bone structures without the use of radiation.

Participants will:

1. Undergo MRI scans of their skeletal system that will then be processed using DL.
2. Undergo CT scans of the same body region for comparison purposes.

ELIGIBILITY:
Inclusion Criteria:

* Referral for a clinically indicated MRI examination of the musculoskeletal system to assess inflammatory and degenerative joint changes.
* Willingness to sign the informed consent form.
* No contraindications for a CT examination (e.g., claustrophobia).

Exclusion Criteria:

* No signed informed consent form.
* Patients under 18 years of age.
* Pregnant women.
* The calculated effective dose of the CT examination exceeds 5 mSv.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Total score for bone erosions | one day (day of MRI and CT examination)
  Each bone is scored separately. The scale is 0-10, based on the proportion of eroded bone compared to the "assessed bone volume," judged on all available images: 0: no erosion; 1: 1-10% of bone eroded; 2: 11-20%, etc. For long bones, the "assessed bone volume" is from the articular surface (or its best estimated position if absent) to a depth of 1 cm, while in carpal/tarsal bones it is the whole bone.
  Example of bone list for hands: carpal bones, distal radius, distal ulna, metacarpal bases; metacarpophalangeal, MCP, joints: metacarpal head, phalangeal base; maximum points: 230.
  A higher score means more bone erosions.
  Note: The total score will vary according to body area imaged, this will be taken into account in the final analysis.
Total score for joint space narrowing | one day (day of MRI and CT examination)
  0: no narrowing, 1: focal or mild (< 33%), 2: moderate (34-66%), 3: moderate to severe (67-99%), 4: ankylosis
  A higher score means more joint space narrowing.
  Note: The total score will vary according to body area imaged, this will be taken into account in the final analysis.
Visibility of cortical bone | one day (day of MRI and CT examination)
  Scale from 1 to 4
  1. hardly visible
  2. diagnostic with some artifact
  3. diagnostic with little artifact
  4. very good depiction
  A higher score means better image quality.
Visibility of trabecular bone | one day (day of MRI and CT examination)
  Scale from 1 to 4
  1. hardly visible
  2. diagnostic with some artifact
  3. diagnostic with little artifact
  4. very good depiction
  A higher score means better image quality.
Visibility of soft tissue calcifications | one day (day of MRI and CT examination)
  Scale from 1 to 4
  1. hardly visible
  2. diagnostic with some artifact
  3. diagnostic with little artifact
  4. very good depiction
  A higher score means better image quality.
Contrast to noise ratio | one day (day of MRI and CT examination)
  Average signal of erosion minus average signal of adjacent healthy bone, divided by the average background signal
  A higher score means better contrast of erosions when standardized for healthy adjacent bone and against the background.
Signal to noise ratio | one day (day of MRI and CT examination)
  Average signal of erosion divided by the average background signal
  A higher score means better contrast of erosions against the background.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No